CLINICAL TRIAL: NCT05096819
Title: Evaluation of the Usefulness of Adopting Remote, Mobile-based 6MWT Among Hospital Outpatients (the 6-APPnow), Within the Constraints Imposed by the SARS-COV2 Pandemic
Acronym: 6-APPnow
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Malmö University (Other)
Responsible Party: Principal Investigator, Elizabeth Orchard, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: PID15408
Record Dates: First submitted 2021-06-05; First posted 2021-10-27 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients Using the 6MWT App in the Community — Patients under the care of the cardiovascular clinics in Oxford, who used the Timed Walk app to perform 6MWT in their community during the CODIV19 pandemic period
Other: Volunteers for 6MWT distance comparison — Volunteers (cardiac patients and hospital staff) who performed 10 6MWT using the TimedWalk app and a trundle wheel simultaneously. Five tests were performed following instructions and 5 were performed introducing errors. Aim is to measure app accuracy under different circumstances.

SUMMARY:
The six-minute walk test (6MWT) is a standard method for measuring exercise capacity in patients with cardiopulmonary disease such as pulmonary hypertension (PAH) and measures how far a patient can walk in 6 minutes. The test is usually performed in the hospital, by walking along a hospital corridor. Since the outbreak of SARS-CoV-2, there has been a need to minimise patient contact with hospitals and their staff to reduce transmission of the virus. In a previous research project called 6APP, the investigators designed, developed and evaluated a mobile phone app, to allow them to perform the 6MWT in the community. Given the current circumstances, cardiovascular outpatients including patients in the PAH clinic at Oxford University Hospitals are being recommended to use an app derived from that project to provide their 6MWT distance to the clinical team for assessment, in addition to their symptoms and general well-being. This is felt to be more appealing to the patients, and would reduce the time spent in hospital on the day of their outpatient appointment. The investigators plan to measure the usefulness of adopting remote, mobile-based 6MWT among hospital outpatients, within the constraints imposed by the SARS-COV2 pandemic.

DETAILED DESCRIPTION:
Context:

Since the outbreak of SARS-CoV-2, health care systems have been subject to increased pressures. This is mainly due to infected patients being admitted to the medical wards and intensive care units, but also due to the requirement to reduce exposure of both healthcare professionals and patients to COVID by minimising contact. There are indications that reduced access to healthcare services during the pandemic is responsible for more than half of excess deaths in the United States. In response to this, the CDC is advocating the use of telemedicine to keep providing a remote version of healthcare services. A study of telemedicine services in China used during COVID-19 pandemic showed that they reduced burden on hospitals, prevented overcrowding, reduced the risk of cross-infection, and relieved patients' anxiety. The use of telemedicine is also being developed in Europe, where many patients are being denied the use of clinical services, like cardiac rehabilitation, because of centres being closed. In the context of the NHS, an increased use of telemedicine services is being observed. The NHS long-term plans do, in fact, include tele-consultations as a pillar for its sustainability. Healthwatch have produced useful advice for outpatient clinicians to consider avoiding asking patients to attend physical outpatient appointments where a clinically-appropriate and accessible alternative exists. Where an appointment is clinically necessary, the national benchmark is that at least 25% could be conducted by telephone or video including 60% of all follow-up appointments. Initial promising results are being seen in the context of diabetes, where virtual clinics are recommended as mitigation to the pandemic.

The 6MWT:

To assess patient's exercise capacity, the six-minute walk test (6MWT) is a standard method used in patients with cardiopulmonary disease such as Heart Failure (HF) or Pulmonary arterial Hypertension (PAH). The 6MWT measures how far a patient can walk in 6 minutes. Walking is an activity performed every day, by most patients except for those most severely limited. By assessing patients' ability to exercise, the 6MWT provides a global assessment of respiratory, cardiovascular, neuromuscular and cognitive function. The 6MWT does not differentiate what limits the patient, nor does it assess maximal exercise capacity. Instead, the 6MWT allows the patient to exercise at a daily functional level, and is a useful tool for assessing changes after a therapeutic intervention, and correlates with a subjective improvement in dyspnoea.

In PAH the 6MWT is used to evaluate patients' response to treatment, with an increase in 6MWT distance of greater than 42 m being considered a clinically significant improvement . Furthermore, change in 6MWT distance correlates with VO2 max, NYHA class and mortality in those patients, providing an objective assessment of disease progression, prognosis and response to treatment. It is a universally accepted test as it is safe and easily performed by the patient.

Cardiovascular outpatient management during the pandemic:

Since the outbreak of SARS-CoV-2, the standard regime of care for outpatients with cardiovascular disease has been affected. For example, in PAH patients, the normal regime of a 6MWT, echocardiogram and face to face consultation was abandoned as those patients were felt to be extremely clinically vulnerable, and therefore were recommended to shield at home. Therefore patients needed to be assessed without having any face to face contact, unless in an emergency. In cardiovascular outpatient clinics in Oxford, patients were regularly contacted by phone to replace face to face visits. During these phone calls, questions about the general status of the patient are asked, i.e. how far they think they can walk and whether they have noticed a change in their exercise capacity or functional capacity, but no objective data, like the results of the 6MWT, were available for assessment.

Telemedicine services for pulmonary hypertension:

In a previous research project called 6APP, we designed, developed and evaluated a mobile-health "app" (a type of telemedicine where patients use their mobile phones), to allow them to perform the 6MWT in the community. We hypothesized that a test conducted by patients, in their environment, would reflect more the patient's functional status, would free up healthcare resources and would be less stressful and costly for the patients themselves.

The app allowed patients to perform the test both indoors, by walking back and forth along a corridor of fixed length, and outdoors, using the localization system (like the GPS). In our study with 30 PAH patients, we proved that the app is accurate when used outdoors, the measurements are reliable and repeatable and the method is well-accepted by patients. After these encouraging results, the app has been simplified and made available for free for both Android and iPhones under the name of "Timed Walk". The original app was developed by Dario Salvi at the Institute of Biomedical Engineering of the Oxford University. The current app, which uses the same validated outdoors test approach, is instead maintained by the Malmo, University Sweden, where Dr. Salvi is currently employed.

Given the circumstances during the pandemic period, the PH clinic in Oxford and other cardiovascular outpatient clinics were recommending patients to use the Timed Walk app, the results of which were being used by the clinical team to assess patients in addition to their symptoms and general well-being. This is felt to be more appealing to the patients, and would reduce the time spent in hospital on the day of their outpatient appointment. The app only allows outdoor tests (as these proved to be more reliable and practical) and to share 6MWT data via email if patients want to.

Goal:

The goal of this study is to contribute to existing research on the adoption of remote mobile-based 6MWT through a mixed methods approach where we mix of complementing quantitative and qualitative data to validate the use of an app within the context of the pandemic.

Methods:

Outpatients undergoing follow up in the cardiovascular outpatient clinics in Oxford, who were able to walk and use a smartphone, were considered eligible. Some of these patients were already using the app, prior to the start of the study, for example in the case of the pulmonary hypertension clinic. Prospective participants were approached by a member of the clinical team for consideration and recruited during their regular outpatient consultation either via phone call or during a visit to the clinic. Participants in the study were asked to download the Timed Walk app and use it to perform a 6MWT in the community, outdoors, at least once a month, and to report the measured 6MWD to the clinicians during the outpatient consultations, via phone or in the clinic.

We did not sample participants as the aim was to involve all patients in the cardiovascular clinics who required a 6MWT and were able to use the app. However, as restrictions started to be lifted in 2022 and practical reasons made the recruitment pace slower than desired (about 4 patients per month), a decision was made to stop recruitment after the 100th patient was selected.

In order to assess the impact the app had on the clinical management of consented patients, at each consultation (either through phone or face to face visit) the clinician who contacted the patient logged any study-related event on a spreadsheet marked with a code, including distance walked during the 6MWT and medical decisions taken. Coding was used to simplify and automate later analysis and was defined in collaboration with the clinical professionals that were part of the study.

As one of the aims of the study was to understand if patients are able and willing to use the app, we used and adapted the broad and validated technology acceptance model for mobile health services and the uMARS questionnaires.

In addition to clinical impact and user acceptance, we wanted to confirm the reliability of the app-based measurements by comparing the 6MWD gathered through the smartphone with a reference. A group of 12 volunteers, patients and staff, were invited after the study period was completed. This included performing 10 6MWT each, using the app and a trundle wheel used as reference simultaneously.

To study the accuracy of the estimated distance under different conditions, participants were instructed to perform 5 tests walking along paths known to obtain the best distance estimation (straight or gently curved paths) and 5 tests walking over paths that are suspected to be more challenging for the app (including narrow curves, U-turns or in confined spaces). We refer to the former type of path as conventional and the latter as unconventional.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in Oxford clinics
* Owning or having access to a smartphone with either Android or iOS
* Being able to use a smartphone app
* Being able to walk

Exclusion Criteria:

* Long term oxygen therapy
* Cognitive impairments
* Cannot use a smartphone
* Pregnancy
* Not able to complete a 6MWT
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients under the care of the cardiovascular clinics in Oxford, who are able to walk and use a smartphone
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Orchard, MA, MBBS, FRCP, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Woolf SH, Chapman DA, Sabo RT, Weinberger DM, Hill L. Excess Deaths From COVID-19 and Other Causes, March-April 2020. JAMA. 2020 Aug 4;324(5):510-513. doi: 10.1001/jama.2020.11787. PMID 32609307
- [Background] Liu L, Gu J, Shao F, Liang X, Yue L, Cheng Q, Zhang L. Application and Preliminary Outcomes of Remote Diagnosis and Treatment During the COVID-19 Outbreak: Retrospective Cohort Study. JMIR Mhealth Uhealth. 2020 Jul 3;8(7):e19417. doi: 10.2196/19417. PMID 32568722
- [Background] Alderwick H, Dixon J. The NHS long term plan. BMJ. 2019 Jan 7;364:l84. doi: 10.1136/bmj.l84. PMID 30617185
- [Background] Quinn LM, Davies MJ, Hadjiconstantinou M. Virtual Consultations and the Role of Technology During the COVID-19 Pandemic for People With Type 2 Diabetes: The UK Perspective. J Med Internet Res. 2020 Aug 28;22(8):e21609. doi: 10.2196/21609. PMID 32716898
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] Gabler NB, French B, Strom BL, Palevsky HI, Taichman DB, Kawut SM, Halpern SD. Validation of 6-minute walk distance as a surrogate end point in pulmonary arterial hypertension trials. Circulation. 2012 Jul 17;126(3):349-56. doi: 10.1161/CIRCULATIONAHA.112.105890. Epub 2012 Jun 13. PMID 22696079
- [Background] Mathai SC, Puhan MA, Lam D, Wise RA. The minimal important difference in the 6-minute walk test for patients with pulmonary arterial hypertension. Am J Respir Crit Care Med. 2012 Sep 1;186(5):428-33. doi: 10.1164/rccm.201203-0480OC. Epub 2012 Jun 21. PMID 22723290
- [Background] Salvi D, Poffley E, Orchard E, Tarassenko L. The Mobile-Based 6-Minute Walk Test: Usability Study and Algorithm Development and Validation. JMIR Mhealth Uhealth. 2020 Jan 3;8(1):e13756. doi: 10.2196/13756. PMID 31899457
- [Background] Stoyanov SR, Hides L, Kavanagh DJ, Wilson H. Development and Validation of the User Version of the Mobile Application Rating Scale (uMARS). JMIR Mhealth Uhealth. 2016 Jun 10;4(2):e72. doi: 10.2196/mhealth.5849. PMID 27287964

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Using the 6MWT App in the Community: Patients invited to use the TimedWalk app to perform 6MWT in the community during the COVID19 pandemic period
- Volunteers for 6MWT Distance Comparison: Volunteers, patients and staff, who performed additional tests to validate the accuracy of the app
Period: Overall Study
Arm/Group | Patients Using the 6MWT App in the Community | Volunteers for 6MWT Distance Comparison
Started | 55 | 12
Completed | 52 | 12
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: demographics not collected from "Volunteers for 6MWT Distance Comparison" Arm
Groups:
- Volunteers for 6MWT Distance Comparison: Demographics data was not collected for this group. Nine of the volunteers were patients involved in the study, three were healthy subjects from the hospital staff.
- Total: Total of all reporting groups
Arm/Group | Patients Using the 6MWT App in the Community | Volunteers for 6MWT Distance Comparison | Total
Number analyzed (Participants) | 55 | 0 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.80 (17.49) |  | 44.80 (17.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 |  | 25
  Male | 30 |  | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Undertaking an App-based 6MWT
Description: Percentage of participants who perform at least one app-based 6MWT per month before patient consultation
Time Frame: At 3, 6, 9 and 12 months after the start of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Using the 6MWT App in the Community
Number analyzed (Participants) | 55
Participants | 24

2. Secondary Outcome: Accuracy of the App-based 6MWT Distance Measurement
Description: Measurement of walked distance (6MWD) measured by the app compared with a trundle wheel reference: conventional tests where users followed instructions (walking on straight paths, avoiding tall structures), unconventional tests where users were free to move as they preferred
Time Frame: 1 year
Population: Difference in 6MWT distance as measured by the app versus as measured by the trundle wheel, used simultaneously
Measure: Mean (Standard Deviation); unit: metre
Units Other Than Participants: Pairs of 6MWT distances (app vs ref)
Groups:
- Volunteers Who Tested the App With a Trundle Wheel: Volunteers, from the patients cohort and staff, that volunteered to perform 10 6MWT with the app the trundle wheel. Five tests were performed following instructions and five were performed in an "unconventional" way.
Arm/Group | Volunteers Who Tested the App With a Trundle Wheel
Number analyzed (Participants) | 12
Number analyzed (Pairs of 6MWT distances (app vs ref)) | 107
metre
  conventional tests | 3.6 (15.8)
  unconventional tests | 73.0 (122.8)
  all tests | 37.4 (92.7)

3. Secondary Outcome: Number and Percentage of Logged Events That Were Triggered by Variations in the App-based 6MWD
Description: Number (and percentage) of clinical investigations and multidisciplinary team discussions (partially) triggered by variations in app-based 6MWD
Time Frame: At 3, 6, 9 and 12 months after the start of the study
Population: Percentage of clinical investigations and multidisciplinary team discussions where variations in app-based 6MWD was a contributing factor
Measure: Count of Units; unit: Logged events
Units Other Than Participants: Logged events
Arm/Group | Patients Using the 6MWT App in the Community
Number analyzed (Participants) | 48
Number analyzed (Logged events) | 51
Logged events | 21

4. Secondary Outcome: Usability and Acceptance of the App
Description: uMARS usability questionnaire and Technology Acceptance questionnaire. Reported average for all dimensions on a 1 to 5 scale with 1 being most negative and 5 being most positive
Time Frame: 12 months
Population: Answers to uMARS questionnaire and Technology Acceptance Model, Likert scale 1 to 5 with 1 being most negative and 5 being most positive
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Patients Using the 6MWT App in the Community
Number analyzed (Participants) | 25
Scores on a scale
  uMARS | 3.89 (0.97)
  TAM | 3.75 (0.97)

5. Secondary Outcome: Comparison of 6MWT During Pandemic and Pre-pandemic
Description: Number of 6MWTs performed during in 2018 in clinic (collected retrospectively, after enrollment), and number of tests performed in 2022 in clinic and with the app, for the same cohort.
Time Frame: 2018 (12 months, retrospectively collected) and 2022 (12 months)
Population: Comparison of a pre-pandemic year (2018) and 2022 in terms of 6MWT performed on the study cohort. The tests in 2022 include the ones performed in clinic and the ones performed with the app.
Measure: Number; unit: 6MWT
Arm/Group | Patients Using the 6MWT App in the Community
Number analyzed (Participants) | 49
6MWT
  2018 at clinic | 17
  2022 at clinic and with app | 600

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Event: any untoward medical occurrence in a participant, including occurrences which are not necessarily caused by or related to the intervention. Mild: awareness of signs or symptoms that does not interfere with the subject's usual activity or is transient that resolved without treatment and with no sequelae. Moderate: a sign or symptom, which interferes with the subject's usual activity. Severe: incapacity with inability to do work or perform usual activities.
Groups:
- Volunteers for 6MWT Distance Comparison: Volunteers who validated the accuracy of the 6MWT app
Arm/Group | Patients Using the 6MWT App in the Community | Volunteers for 6MWT Distance Comparison
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/12
Other Adverse Events (participants affected / at risk) | 0/55 | 0/12

LIMITATIONS AND CAVEATS:
The study did not employ a control group, therefore it is impossible to ascertain if patients would have received the same level of care without the use of the app.

This study was conducted under special circumstances due to the restrictions imposed during the COVID 19 pandemic. In that period patients may have been keener to use telemedicine to ensure they were being followed up. The results obtained may therefore not generalize outside of those circumstances.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT05096819/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT05096819/ICF_001.pdf